CLINICAL TRIAL: NCT04615871
Title: Semaglutide to Reduce Myocardial Injury in PATIents With COVID-19 Randomized Controlled Trial
Brief Title: Semaglutide to Reduce Myocardial Injury in PATIents With COVID-19
Acronym: SEMPATICO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vladimír Džavík (Other)
Collaborators: Unity Health Toronto (Other); Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Vladimír Džavík, Principal Investigator, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHNSEMPATICO1
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Covid19; Myocardial Injury
Keywords: Covid-19; myocardial injury; GLP-1 agonist; semaglutide
MeSH Terms: conditions — COVID-19 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive active treatment - s.c. semaglutide for 4 weekly doses in addition to standard of care or control - standard of care only
Who Masked: Outcomes Assessor
Masking Description: Randomized open-label blinded evaluation trial. There will be an independent events adjudication committee
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- semaglutide (Experimental): Eligible subjects randomized to this arm will receive semaglutide 0.25 mg s.c. after randomization (Day 0), then semaglutide 0.5 mg s.c. on Day 7, Day 14 and Day 21 in addition to standard of care.
  Interventions: Drug: semaglutide
- control (No Intervention): Eligible subjects randomized to the control arm will receive no active treatment, only standard of care.

INTERVENTIONS:
Drug: semaglutide — semaglutide 0.25 mg s.c. on Day 0 after randomization, then semaglutide 0.5 mg s.c. on Day 7, Day 14 and Day 21
  Other Names: Ozempic
  Arms: semaglutide

SUMMARY:
With the results of this study the investigators aim to identify an effective treatment that will reduce morbidity and mortality of patients with symptomatic COVID-19 infection, which would in turn reduce the burden on the healthcare system by decreasing the need for intensive care.

Objectives: The main objective of this research is to determine if once weekly treatment with the GLP-1 agonist semaglutide for 4 doses will reduce cardiac as well as non-cardiac complications of COVID-19 infection.

Study Plan: The study design is prospective randomized open-label blinded-evaluation (PROBE). Eligible patients with symptomatic COVID-19 infection and an enhanced risk profile as described above, who have been admitted to hospital due to symptoms of COVID-19 infection but do not as yet require critical care will be approached to participate in this study. Provided there are no exclusion criteria and the participants agree by means of documented written informed consent, The participants the participants will be randomized to receive s.c. semaglutide 0.25 mg s.c. or control immediately after randomization and then 0.5 mg s.c. at Day 7, Day 14 and Day 21. Blood will be drawn at Day 7±2 and Day 14±2 for the cardiac troponin biomarker and safety parameters. ECG will be obtained at Day 7±2 and Day 14±2. Primary outcome will be assessed on Day 28.

Primary outcome measure: A composite of (1) death from any cause or (2) mechanical ventilation (invasive or non-invasive) at 28 days.

Major secondary outcome measure:

(1) an elevation to >99th percentile URL upper reference limit (URL) in those with a baseline cardiac troponin level ≤99th percentile URL; or 3x elevation from baseline in those with a baseline cardiac troponin >99th percentile URL; measured at 1 week (7-days) post randomization.

Other major secondary outcome measure:

A composite of

1. Death from any cause, mechanical ventilation or vasopressor or ECLS support at 28 days
2. an elevation to >99th percentile URL in those with a normal baseline troponin level; or 3x elevation from baseline in those with a baseline troponin; measured at 1 and 2 weeks (7±2 and 14±2 days) post randomization.

DETAILED DESCRIPTION:
6.1 Background

The current COVID-19 pandemic is rapidly spreading with a global total of ~35 million cases, with close to 170,000 cases and over 9,500 deaths in Canada alone (as of 10/05/2020). Most affected patients have mild or even no symptoms, however, those requiring hospitalization have a more severe presentation including pneumonia, acute respiratory distress syndrome (ARDS), cardiovascular collapse and death. There is mounting evidence that myocardial injury, occurring in 8-28% of hospitalized patients, has a major impact on mortality. In a study from Wuhan in China, mortality was 59.6% in COVID-19 patients with an elevated troponin and only 8.9% in those with a normal troponin level. ARDS was also more common in troponin-positive patients. The pathophysiology of myocardial injury following COVID-19 infection is not well understood, but may include viral myocarditis, cardiomyocyte injury from systemic cytokine storm, reductions in myocardial blood flow from micro- and macro-vascular thromboses, and severe hypoxemia in the setting of pre-existing cardiovascular disease (CVD).1 Higher rates of adverse outcomes with COVID-19 have also been noted in patients with hypertension and diabetes. Based on these data, approaches to prevent or reduce the vascular consequences of COVID-19 may be beneficial and should be prioritized for rapid evaluation in controlled clinical trials.

Currently there is a paucity of approved therapies for COVID-19 infection. Current interventions are either supportive in nature or experimental anti-viral, anti-inflammatory, or anti-coagulant in nature. Only dexamethasone has recently been shown to reduce mortality. To date, there is no proposed treatment directly addressing the mechanisms of increased cardiovascular risk in this deadly disease. The investigators have strong rationale and world-leading expertise in this area. This is a prospective, randomized, controlled, open-label, blinded-evaluation, exploratory (vanguard) study in hospitalized symptomatic COVID-19 patients age with any two of the following high-risk features: age >60 years, obesity (BMI> 30), diabetes (by history - with or without medical treatment), hypertension (on any treatment), cardiovascular disease (by history), chronic kidney disease (eGFR <60) or elevated biomarkers on admission to hospital (troponin, d-dimer). Eligible and consented patients will be randomized to one of the following two treatment regimens in a 1:1 ratio: (1) semaglutide 0.25 mg s.c. immediately after randomization at baseline, then 0.5 mg s.c. at day 7, day 14, and day 21. The end of treatment period and primary outcome assessments will occur on day 28. Final secondary clinical outcome assessment will be at 180 days.

With the results of this study the investigators aim to identify an effective treatment that will reduce morbidity and mortality of patients with symptomatic COVID-19 infection, which would in turn reduce the burden on the healthcare system by decreasing the need for intensive care.

Objectives: The main objective of this research is to determine if once weekly treatment with the GLP-1 agonist semaglutide for 4 doses will reduce cardiac as well as non-cardiac complications of COVID-19 infection.

Study Plan: The study design is prospective randomized open-label blinded-evaluation (PROBE). Eligible patients with symptomatic COVID-19 infection and an enhanced risk profile as described above, who have been admitted to hospital due to symptoms of COVID-19 infection but do not as yet require critical care will be approached to participate in this study. Provided there are no exclusion criteria and the participants agree by means of documented written informed consent, The participants will be randomized to receive s.c. semaglutide 0.25 mg s.c. or control immediately after randomization and then 0.5 mg s.c. at Day 7, Day 14 and Day 21. Blood will be drawn at Day 7 and Day 14 for the cardiac troponin biomarker and safety parameters. ECG will be obtained at Day 7±2 and Day 14±2. Primary outcome will be assessed on Day 28.

Primary outcome measure: A composite on Day 28 after randomization of (1) death from any cause, (2) mechanical ventilation (invasive or non-invasive [bilevel positive airway pressure or BIPAP])

Major secondary outcome measure:

(1) an elevation to >99th percentile URL upper reference limit (URL) in those with a baseline cardiac troponin level ≤99th percentile URL; or 3x elevation from baseline in those with a baseline cardiac troponin >99th percentile URL; measured at Day 7±2 and Day 14±2 post randomization.

Other major secondary outcome measure:

1. A composite on Day 28 after randomization of (1) death from any cause, (2) mechanical ventilation (invasive or non-invasive [bilevel positive airway pressure] (3) an elevation to >99th percentile URL in those with a normal baseline troponin level; or 3x elevation from baseline in those with a baseline troponin; measured at Day 7±2 and Day 14±2 post randomization.
2. ECG at Day 7±2 and Day 14±2: QRS and ST-T wave changes
3. 28-day organ support-free days
4. A composite of death or intensification of medical therapy in hospitalized symptomatic patients infected with the COVID-19 virus, that includes the need for ECLS, mechanical ventilation (invasive or non-invasive [BIPAP]) and/or vasopressor/inotropic therapy on Day 180 post randomization.

Sample size estimation: The study plan is to enroll 50 patients in an initial feasibility phase and continue to a total of 400 patients in the complete vanguard study based on the assumption of a 20% primary event rate in the control group, and a 50% relative risk reduction in the event rate in the active treatment arm. The rationale for the large effect size to be tested is the need for a rapid answer for this life-threatening pandemic. A conditional power analysis will allow the investigators to adjust the study size as needed. When 70% of the randomized patients have reached the 28-day time-point, conditional power will be estimated on the primary outcome. If the conditional power is between 60% and 80%, the sample size will be adjusted to raise the power to 80%.

Planned subgroup analyses: Planned subgroup analyses for the primary endpoint include: 1) Diabetes vs. no diabetes, 2) baseline troponin >99% percentile URL vs. not, 3) age < 60 y vs. age ≥ 60 y, 4) eGFR < 60 mL/min vs. eGFR ≥ 60 mL/min, , 6) male vs. female. These subgroup effects will be explored using a treatment-interaction test.

ELIGIBILITY:
Inclusion Criteria:

Symptomatic* COVID-2 infection confirmed by a positive COVID-19 test requiring hospitalization [or equivalent health care setting] with any two of the following high-risk features:

* age ≥ 60 years
* obesity (BMI >30)
* diabetes mellitus
* hypertension (on treatment or recently diagnosed)h
* coronary artery, cerebrovascular or peripheral vascular disease∫
* chronic kidney disease (CKD) [eGFR <60 mL/min/1.73m2 using the CKD Epidemiology Collaboration equation
* admission troponin >99% of ULN
* admission d-dimer > 1µg/ml
* O2 saturation ≤93% e on room air or need for any O2 therapy

Exclusion Criteria:

* Age <18 years
* History of pancreatitis
* History of multiple endocrine neoplasia or medullary thyroid cancer
* Current use of a GLP-1 receptor agonist [use of a DPP-4 inhibitor is allowed]
* Positive beta-HCG (pregnancy test is mandated with baseline bloodwork for all female subjects ≤50 years of age
* Breastfeeding, if they intend to continue breastfeeding
* Elevation of serum lipase, direct (conjugated) bilirubin, or alkaline phosphatase (ALP) more than 3X the upper limit of normal on baseline bloodwork
* history of decompensated heart failure with reduced ejection fraction (<35%) within 90 days, or known stable NYHA class IV heart failure prior to their COVID-19 illness
* imminent mechanical ventilation or death
* O2 therapy with high flow nasal cannula at FiO2 >50% or already on mechanical ventilation
* Any marker of hemodynamic instability at baseline defined as persistent SBP <90 mmHg after rehydration, or > 220 mmHg after receiving routine antihypertensive therapy, or HR <50 bpm or > 140 bpm after rehydration.
* inability to provide informed consent from patient or Substitute Decision Maker (SDM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Composite of death or mechanical ventilation | 28 days after randomization
  All cause death or invasive or non-invasive mechanical ventilation

SECONDARY OUTCOMES:
cardiac troponin level | 7±2 days after randomization
  (1) an elevation to >99th percentile URL upper reference limit (URL) in those with a baseline cardiac troponin level ≤99th percentile URL; or 3x elevation from baseline in those with a baseline cardiac troponin >99th percentile URL; measured at 1 week (7-days) post randomization.
cardiac troponin level | 14±2 days after randomization
  (1) an elevation to >99th percentile URL upper reference limit (URL) in those with a baseline cardiac troponin level ≤99th percentile URL; or 3x elevation from baseline in those with a baseline cardiac troponin >99th percentile URL; measured at 1 week (7-days) post randomization.
ECG | Day 7±2 and Day 14±2
  The ECG will be evaluated for deviation from normal or from baseline (QRS, ST-T wave changes
28-day organ support-free days | 28 days
  The number of days that a patient is alive and free of organ support through 28 days after trial entry. Organ support is defined by receipt for non-invasive mechanical ventilation, high flow nasal cannula oxygen, mechanical ventilation, or vasopressor therapy.
  Non-invasive mechanical ventilation is defined as bilevel positive airway pressure (BIPAP) or continuous positive airway pressure (CPAP) when used for acute respiratory support (Use of BIPAP or CPAP at night or when sleeping for sleep apnea is not considered organ support) High Flow Nasal Cannula Oxygen: defined as receiving ≥30 l/min flow at FiO2 ≥40% Invasive mechanical ventilation is defined as positive pressure ventilation through endotracheal tube or tracheostomy Vasopressor support includes infusion of any vasoactive or inotropic medication
A composite of death or intensification of medical therapy | 180 days
  Intensification of medical therapy includes the need for ECLS, mechanical ventilation (invasive or non-invasive [BIPAP]) and/or vasopressor/inotropic therapy on Day 180 post randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Dzavik, MD, Principal Investigator — University Health Network, Toronto; Mansoor Husain, MD, Principal Investigator — University Health Network, Toronto
Locations (10):
- Brazil (2):
  - Instituto Prevent Senior, São Paulo
  - State University of Campinas, São Paulo
- Canada (4):
  - Trillium Health Partners, Mississauga, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network - Peter Munk Cardiac Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Mexico (3):
  - Hospital de Infectologia, Mexico City
  - Hospital General Regional, Mexico City
  - Hospital Regional 2, Querétaro
- Sandwell and West Birmingham NHS Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No